CLINICAL TRIAL: NCT01233258
Title: A Phase II/III, Randomized, Cross-over, Open-label Trial to Demonstrate Superiority of Prophylaxis Over On-demand Therapy in Previously Treated Subjects With Severe Hemophilia A Treated With Plasma Protein-free Recombinant FVIII Formulated With Sucrose (BAY 81-8973)
Brief Title: A Trial to Compare Prophylaxis Therapy to On-demand Therapy With a New Full Length Recombinant FVIII in Patients With Severe Hemophilia A
Acronym: Leopold II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14319; 2009-012150-20 (EudraCT Number)
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Hemophilia A
Keywords: Haemophilia treatment; rFVIII
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1: rFVIII on demand first CS/EP then CS/ADJ (Experimental): Participants received on-demand treatment with recombinant factor VIII (rFVIII, BAY81-8973) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months, followed by cross-over to study drug assayed by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months.
  Interventions: Biological: rFVIII (BAY81-8973) on demand
- Arm 2: rFVIII on demand first CS/ADJ then CS/EP (Experimental): Participants received on-demand treatment with rFVIII (BAY81-8973) assayed by CS/ADJ for 6 months, followed by cross-over to study drug assayed by CS/EP for 6 months.
  Interventions: Biological: rFVIII (BAY81-8973) on demand
- Arm 3: rFVIII prophylaxis low-dose first CS/EP then CS/ADJ (Experimental): Participants received low dose prophylaxis treatment at 20, 25 or 30 IU/kg twice per week with rFVIII(BAY81-8973) measured by CS/ EP for 6 months then crossed over to study drug measured by CS/ADJ for 6 months.
  Interventions: Biological: rFVIII (BAY81-8973) prophylaxis low-dose
- Arm 4: rFVIII prophylaxis low-dose first CS/ADJ then CS/EP (Experimental): Participants received low dose prophylaxis treatment at 20, 25 or 30 IU/kg twice per week with rFVIII (BAY81-8973) measured by CS/ADJ for 6 months then crossed over to study drug measured by CS/ EP for 6 months.
  Interventions: Biological: rFVIII (BAY81-8973) prophylaxis low-dose
- Arm 5: rFVIII prophylaxis high-dose first CS/EP then CS/ADJ (Experimental): Participants received high dose prophylaxis treatment at 30, 35 or 40 IU/kg 3 times per week with rFVIII (BAY81-8973) measured by CS/ EP for 6 months then crossed over to study drug measured by CS/ADJ for 6 months.
  Interventions: Biological: rFVIII (BAY81-8973) prophylaxis high-dose
- Arm 6: rFVIII prophylaxis high-dose first CS/ADJ then CS/EP (Experimental): Participants received high dose prophylaxis treatment at 30, 35 or 40 IU/kg 3 times per week with rFVIII(BAY81-8973) measured by CS/ADJ for 6 months then crossed over to study drug measured by CS/ EP for 6 months.
  Interventions: Biological: rFVIII (BAY81-8973) prophylaxis high-dose

INTERVENTIONS:
Biological: rFVIII (BAY81-8973) on demand — Participants received on-demand treatment with rFVIII (BAY81-8973) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months and by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months, sequence according to randomization
  Arms: Arm 1: rFVIII on demand first CS/EP then CS/ADJ; Arm 2: rFVIII on demand first CS/ADJ then CS/EP
Biological: rFVIII (BAY81-8973) prophylaxis low-dose — Participants received low dose prophylaxis treatment at 20, 25 or 30 IU/kg twice per week with rFVIII (BAY81-8973) assayed by CS/EP for 6 months and by CS/ADJ for 6 months, sequence according to randomization.
  Arms: Arm 3: rFVIII prophylaxis low-dose first CS/EP then CS/ADJ; Arm 4: rFVIII prophylaxis low-dose first CS/ADJ then CS/EP
Biological: rFVIII (BAY81-8973) prophylaxis high-dose — Participants received high dose prophylaxis treatment at 30, 35 or 40 IU/kg 3 times per week with rFVIII (BAY81-8973) assayed by CS/EP for 6 months and by CS/ADJ for 6 months, sequence according to randomization.
  Arms: Arm 5: rFVIII prophylaxis high-dose first CS/EP then CS/ADJ; Arm 6: rFVIII prophylaxis high-dose first CS/ADJ then CS/EP

SUMMARY:
The objective of the trial is to demonstrate that 2-3 times per week prophylaxis therapy with BAY81-8973 is superior to on-demand therapy with BAY81-8973 in patients with severe Hemophilia A. The hypothesis is that prophylaxis will result in fewer bleeds than on-demand treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 12 to 65 years
* Severe hemophilia A
* History of more than 150 exposure days (ED) with clotting factor concentrates
* Currently receiving episodic treatment with FVIII; no regular prophylaxis for more than 6 consecutive months in the past 5 years
* No current Factor VIII inhibitor or history of inhibitor
* Willing to use electronic patient diary

Exclusion Criteria:

* Presence of another bleeding disease that is different from hemophilia A
* Thrombocytopenia
* Abnormal renal function
* Presence of active liver disease
* Known hypersensitivity to FVIII

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (45):
- United States (2):
  - Dayton, Ohio
  - Houston, Texas
- Argentina (3):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Corrientes, Corrientes Province
  - Rosario, Santa Fe Province
- China (5):
  - Guangzhou, Guangdong
  - Suzhou, Jiangsu
  - Beijing
  - Shanghai
  - Tianjin
- Colombia (2):
  - Bogotá, Bogota D.C.
  - Bucaramanga, Santander Department
- Olomouc, Czechia
- Hyderabad, India
- Jakarta, Indonesia
- Japan (5):
  - Hiroshima, Hiroshima
  - Nishinomiya, Hyōgo
  - Kashihara, Nara
  - Shinjuku-ku, Tokyo
  - Suginami, Tokyo
- Mexico (2):
  - Guadalajara, Jalisco
  - San Luis Potosí City, San Luis Potosí
- Romania (3):
  - Timișoara, Timiș County
  - Baia Mare
  - Bucharest
- Russia (4):
  - Barnaul
  - Khabarovsk
  - Saint Petersburg
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- Bratislava, Slovakia
- South Africa (2):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
- Taiwan (2):
  - Taichung
  - Taipei
- Bangkok, Thailand, Thailand
- Turkey (Türkiye) (3):
  - Adana
  - Antalya
  - Izmir
- Ukraine (3):
  - Kiev
  - Lviv
  - Simferopol

REFERENCES:
- [Result] Kitchen S, Katterle Y, Beckmann H, Maas Enriquez M. Chromogenic assay for BAY 81-8973 potency assignment has no impact on clinical outcome or monitoring in patient samples. J Thromb Haemost. 2016 Jun;14(6):1192-9. doi: 10.1111/jth.13322. Epub 2016 May 3. PMID 27002680
- [Result] Oldenburg J, Windyga J, Hampton K, Lalezari S, Tseneklidou-Stoeter D, Beckmann H, Maas Enriquez M. Safety and efficacy of BAY 81-8973 for surgery in previously treated patients with haemophilia A: results of the LEOPOLD clinical trial programme. Haemophilia. 2016 May;22(3):349-53. doi: 10.1111/hae.12839. Epub 2016 Mar 1. PMID 26931631
- [Derived] Kavakli K, Yang R, Rusen L, Beckmann H, Tseneklidou-Stoeter D, Maas Enriquez M; LEOPOLD II Study Investigators. Prophylaxis vs. on-demand treatment with BAY 81-8973, a full-length plasma protein-free recombinant factor VIII product: results from a randomized trial (LEOPOLD II). J Thromb Haemost. 2015 Mar;13(3):360-9. doi: 10.1111/jth.12828. PMID 25546368
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from specialized hemophilia treatment centers.
Pre-assignment Details: 83 participants were randomized, but 3 of these terminated the study before their first injection of study drug.
Groups:
- On Demand, BAY 81-8973 Potency First EP Then ADJ: Participants received on-demand treatment with recombinant factor VIII (rFVIII, BAY81-8973) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months, followed by cross-over to study drug assayed by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months.
- On Demand, BAY 81-8973 Potency First ADJ Then EP: Participants received on-demand treatment with rFVIII (BAY81-8973) assayed by CS/ADJ for 6 months, followed by cross-over to study drug assayed by CS/EP for 6 months.
- Low Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ: Participants received low dose prophylaxis treatment at 20, 25 or 30 IU/kg twice per week with rFVIII(BAY81-8973) measured by CS/ EP for 6 months then crossed over to study drug measured by CS/ADJ for 6 months.
- Low Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP: Participants received low dose prophylaxis treatment at 20, 25 or 30 IU/kg twice per week with rFVIII (BAY81-8973) measured by CS/ADJ for 6 months then crossed over to study drug measured by CS/ EP for 6 months.
- High Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ: Participants received high dose prophylaxis treatment at 30, 35 or 40 IU/kg 3 times per week with rFVIII (BAY81-8973) measured by CS/ EP for 6 months then crossed over to study drug measured by CS/ADJ for 6 months.
- High Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP: Participants received high dose prophylaxis treatment at 30, 35 or 40 IU/kg 3 times per week with rFVIII(BAY81-8973) measured by CS/ADJ for 6 months then crossed over to study drug measured by CS/ EP for 6 months.
Period: First Intervention (6 Months)
Arm/Group | On Demand, BAY 81-8973 Potency First EP Then ADJ | On Demand, BAY 81-8973 Potency First ADJ Then EP | Low Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ | Low Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP | High Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ | High Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP
Started | 11 | 10 | 14 | 16 | 16 | 16
Participants Received Treatment | 11 | 10 | 13 | 15 | 16 | 15
Completed | 10 | 10 | 13 | 15 | 16 | 15
Not Completed | 1 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-compliance with study medication | 1 | 0 | 0 | 0 | 0 | 0
Period: Washout (2-3 Days)
Arm/Group | On Demand, BAY 81-8973 Potency First EP Then ADJ | On Demand, BAY 81-8973 Potency First ADJ Then EP | Low Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ | Low Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP | High Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ | High Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP
Started | 10 | 10 | 13 | 15 | 16 | 15
Completed | 10 | 10 | 13 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (6 Months)
Arm/Group | On Demand, BAY 81-8973 Potency First EP Then ADJ | On Demand, BAY 81-8973 Potency First ADJ Then EP | Low Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ | Low Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP | High Dose Prophylaxis, BAY 81-8973 Potency First EP Then ADJ | High Dose Prophylaxis, BAY 81-8973 Potency First ADJ Then EP
Started | 10 | 10 | 13 | 15 | 16 | 15
Completed | 10 | 10 | 13 | 15 | 16 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rFVIII (BAY81-8973) on Demand | rFVIII (BAY81-8973) Prophylaxis Low-dose | rFVIII (BAY81-8973) Prophylaxis High-dose | Total
Number analyzed (Participants) | 21 | 28 | 31 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (10.9) | 28.8 (10.9) | 29.1 (11.5) | 29.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 21 | 28 | 31 | 80

OUTCOME MEASURES:

1. Primary Outcome: Annualized Number of All Bleeds
Description: The annualized number of bleeds experienced by participants
Time Frame: Up to 12 months (6 months per mode of potency assignment according to the randomized cross-over design)
Population: ITT (Intent to Treat). Low and high dose prophylaxis arms and both potencies combined as planned for the statistical analysis to achieve intended sample size.
Measure: Mean (Standard Deviation); unit: Bleeds per year per participant
Groups:
- rFVIII (BAY81-8973) on Demand: Participants received on-demand treatment rFVIII (BAY81-8973) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months and by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months, sequence according to randomization
- rFVIII (BAY81-8973) Prophylaxis Treatment: Participants received prophylaxis treatment with rFVIII (BAY81-8973) at low-dose (20, 25 or 30 IU/kg twice per week ) and high-dose (30, 35 or 40 IU/kg 3 times per week ) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months and by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months, sequence according to randomization.
Arm/Group | rFVIII (BAY81-8973) on Demand | rFVIII (BAY81-8973) Prophylaxis Treatment
Number analyzed (Participants) | 21 | 59
Bleeds per year per participant | 57.7 (24.6) [41.7 to 76.3] | 4.9 (6.8) [0.0 to 7.0]
Statistical Analysis 1: Comparison: rFVIII (BAY81-8973) on Demand vs rFVIII (BAY81-8973) Prophylaxis Treatment; Null hypothesis: bleeding rates are equal, alternative hypothesis rates are unequal. Power calculation: Assumption 5 bleeds per year on prophylactic treatment, 15 on on-demand treatment; 2-sided alpha 5% and 90% power; Test type: Superiority or Other; p = 0.0001, ANOVA — No multiplicity adjustment as only 1 primary endpoint; No adjustment, no transformation of data seemed to be necessary

2. Secondary Outcome: Annualized Number of All Bleeds During CS/EP Period
Description: The annualized number of bleeds experienced by participants while they were taking rFVIII (BAY81-8973) assayed by CS/EP
Time Frame: Up to 6 months (6 months on CS/EP potency assignment)
Population: ITT. Low and high dose prophylaxis arms combined as planned for the statistical analysis to achieve sufficient sample size.
Measure: Mean (Standard Deviation); unit: Bleeds per year per participant
Groups:
- rFVIII (BAY81-8973) on Demand Assayed by CS/EP: Participants received on-demand treatment with rFVIII (BAY81-8973) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months
- rFVIII (BAY81-8973) Prophylaxis Treatment Assayed by CS/EP: Participants received prophylaxis treatment with rFVIII (BAY81-8973) at low-dose (20, 25 or 30 IU/kg twice per week ) and high-dose (30, 35 or 40 IU/kg 3 times per week ) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months.
Arm/Group | rFVIII (BAY81-8973) on Demand Assayed by CS/EP | rFVIII (BAY81-8973) Prophylaxis Treatment Assayed by CS/EP
Number analyzed (Participants) | 21 | 59
Bleeds per year per participant | 57.6 (24.3) [39.4 to 72.7] | 5.1 (8.0) [0.0 to 6.8]
Statistical Analysis 1: Comparison: rFVIII (BAY81-8973) on Demand Assayed by CS/EP vs rFVIII (BAY81-8973) Prophylaxis Treatment Assayed by CS/EP; Null hypothesis: bleeding rates are equal, alternative hypothesis rates are unequal. Power calculation not done for this comparison as not primary comparison; Test type: Superiority or Other; p = 0.0001, ANOVA — No multiplicity adjustment as this is not primary endpoint; No adjustment, no transformation of data seemed to be necessary

3. Secondary Outcome: Annualized Number of All Bleeds During CS/ADJ Period
Description: The annualized number of bleeds experienced by participants while they were taking rFVIII (BAY81-8973) assayed by CS/ADJ
Time Frame: Up to 6 months (6 months on CS/ADJ potency assignment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Bleeds per year per participant
Groups:
- rFVIII (BAY81-8973) on Demand Assayed by CS/ADJ: Participants received on-demand treatment with rFVIII (BAY81-8973) assayed by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months
- rFVIII (BAY81-8973) Prophylaxis Treatment Assayed by CS/ADJ: Participants received prophylaxis treatment with rFVIII (BAY81-8973) at low-dose (20, 25 or 30 IU/kg twice per week ) and high-dose (30, 35 or 40 IU/kg 3 times per week ) assayed by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months
Arm/Group | rFVIII (BAY81-8973) on Demand Assayed by CS/ADJ | rFVIII (BAY81-8973) Prophylaxis Treatment Assayed by CS/ADJ
Number analyzed (Participants) | 20 | 59
Bleeds per year per participant | 59.7 (25.1) [41.0 to 77.8] | 4.8 (6.8) [0.0 to 7.8]
Statistical Analysis 1: Comparison: rFVIII (BAY81-8973) on Demand Assayed by CS/ADJ vs rFVIII (BAY81-8973) Prophylaxis Treatment Assayed by CS/ADJ; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANOVA; No adjustment, no transformation of data seemed to be necessary

4. Secondary Outcome: Percentage of Bleeds Per Participant Controlled With ≤ 2 Injections in Participants Treated on Demand With rFVIII (BAY81-8973)
Description: The percentage of bleeds per participant on on-demand treatment that stopped after two or fewer injections
Time Frame: Up to 12 months (6 months per mode of potency assignment according to the randomized cross-over design)
Population: ITT
Measure: Median (Full Range); unit: Percentage of bleeds
Arm/Group | rFVIII (BAY81-8973) on Demand Assayed by CS/EP | rFVIII (BAY81-8973) on Demand Assayed by CS/ADJ
Number analyzed (Participants) | 21 | 20
Percentage of bleeds | 96.8 [77.8 to 100.0] | 100.0 [65.7 to 100.0]
Statistical Analysis 1: Comparison: rFVIII (BAY81-8973) on Demand Assayed by CS/EP vs rFVIII (BAY81-8973) on Demand Assayed by CS/ADJ; Null hypothesis: the proportion of bleeds controlled by no more than 2 infusions in the CS/EP group plus 10% is less than the proportion of bleeds controlled by no more than 2 infusions in the CS/ADJ group. Alternative hypothesis: the proportion of bleeds controlled by no more than 2 infusions in the CS/EP group plus 10% is greater than or equal to the proportion of bleeds controlled by no more than 2 infusions in the CS/ADJ group. No power calculation since this is not the primary comparison; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 10%; p = 0.0001, Exact Permutation Test for paired sample — No multiplicity adjustment as not primary endpoint; Median Difference (Net) = -0.0001, 95% CI 1-sided [lower limit -0.0490] — Confidence interval calculated with exact Hodges- Lehmann estimates for CS/EP minus CS/ADJ

5. Other Pre Specified Outcome: Number of Bleeds During Treatment
Description: The number of bleeds experienced by each participant
Time Frame: 12 months
Population: ITT
Measure: Median (Inter-Quartile Range); unit: Bleeds
Groups:
- rFVIII (BAY81-8973) Prophylaxis Low-dose: Participants received prophylaxis treatment with rFVIII (BAY81-8973) at low-dose (20, 25 or 30 IU/kg twice per week) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months and by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months, sequence according to randomization
- rFVIII (BAY81-8973) Prophylaxis High-dose: Participants received prophylaxis treatment with rFVIII (BAY81-8973) at high-dose (30, 35 or 40 IU/kg 3 times per week) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months and by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months, sequence according to randomization
Arm/Group | rFVIII (BAY81-8973) on Demand | rFVIII (BAY81-8973) Prophylaxis Low-dose | rFVIII (BAY81-8973) Prophylaxis High-dose
Number analyzed (Participants) | 21 | 28 | 31
Bleeds | 60.0 [42.0 to 77.0] | 4.0 [0.0 to 8.0] | 2.0 [0.0 to 5.0]

6. Other Pre Specified Outcome: Number of Participants With Inhibitory Antibody Formation
Description: A test to ensure that participants have not developed antibodies that will interfere with the action of rFVIII (BAY81-8973)
Time Frame: 3, 6, 9 and 12 months after baseline
Population: Safety population
Measure: Number; unit: Participants
Groups:
- rFVIII (BAY81-8973) Prophylaxis High-dose: Participants received prophylaxis treatment with rFVIII (BAY81-8973) at high-dose (30, 35 or 40 IU/kg 3 times per week ) assayed by CS/EP (Chromogenic Substrate Assay per European Pharmacopoeia) for 6 months and by CS/ADJ (Chromogenic Substrate Assay/label adjusted to one-stage assay) for 6 months, sequence according to randomization.
Arm/Group | rFVIII (BAY81-8973) on Demand | rFVIII (BAY81-8973) Prophylaxis Low-dose | rFVIII (BAY81-8973) Prophylaxis High-dose
Number analyzed (Participants) | 21 | 28 | 31
Participants
  3 months after baseline | 0 | 0 | 0
  6 months after baseline | 0 | 0 | 0
  9 months after baseline | 0 | 0 | 0
  12 months after baseline | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event data reported here were collected from start of first treatment up to 12.5 months (end of observation period).
Description: Abbreviations used in the Adverse Events section: Medical Dictionary for Regulatory Activities (MedDRA)
Groups:
- rFVIII (BAY81-8973) Treatment: Participants received on-demand or prophylaxis treatment with recombinant factor VIII (rFVIII, BAY81-8973) assayed by CS/EP for 6 months and by CS/ADJ for 6 months, sequence according to randomization
Arm/Group | rFVIII (BAY81-8973) Treatment
Serious Adverse Events (participants affected / at risk) | 2/80
Other Adverse Events (participants affected / at risk) | 23/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIII (BAY81-8973) Treatment (N=80)
Head injury (Injury, poisoning and procedural complications) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIII (BAY81-8973) Treatment (N=80)
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 6
Headache (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days